CLINICAL TRIAL: NCT05215951
Title: The Efficacy and Safety of Osimertinib With Platinum Plus Pemetrexed Chemotherapy as First-line Treatment in Advanced Non-small Cell Lung Cancer Patients With Uncommon Epidermal Growth Factor Receptor Mutations: A phase2, Open Label, Single Arm, Multicenter, Exploratory Study
Brief Title: Osimertinib Plus Chemotherapy in Uncommon EGFRm NSCLC
Acronym: MINOVA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment delay study timeline seriously.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5161C00017
Record Dates: First submitted 2021-11-15; First posted 2022-01-31 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib plus standard chemotherapy (Experimental): single-arm
  Interventions: Drug: osimertinib

INTERVENTIONS:
Drug: osimertinib — Dose Formulation: tablet； Dosage Level(s): osimertinib 80 mg QD for oral administration; Dosage formulation, dose reduction:40 mg QD for oral administration
  Other Names: AZD9291; Tagrisso

SUMMARY:
This is an open-label, single-arm, multicenter, exploratory Phase II study sponsored by Astrazeneca Investment (China) Co., LTD. to evaluate the efficacy and safety of Osimertinib with Platinum plus Pemetrexed Chemotherapy, as First-line Treatment in Recurrent or Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Patients with Uncommon Epidermal Growth Factor Receptor Mutations (EGFRm).

DETAILED DESCRIPTION:
Participants successfully enrolled into the study will receive 80mg osimertinib QD p.o. plus standard chemotherapy composed of cisplatin or carboplatin and pemetrexed i.v. on Day 1 of a 21 day cycle (every 3 weeks) for 4 to 6 cycles, followed by osimertinib 80 mg QD p.o. plus pemetrexed maintenance i.v. every 3 weeks until RECIST 1.1-defined radiological progression as judged by the investigator.

Tumour assessments will be performed as per RECISTv1.1 criteria, using computed tomography (CT)/magnetic resonance imaging (MRI). The baseline assessment is part of the screening procedures and should be performed before the start of study intervention.

safety will be assessed in the whole treatment period as well as 28 days after study drug termination for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Provision of signed and dated, written informed consent form prior to any mandatory study-specific procedures, sampling, and analyses.
3. Male or female, at least 18 years of age.
4. Pathologically confirmed nonsquamous NSCLC.
5. Newly diagnosed locally advanced (clinical stage IIIB, IIIC) or metastatic NSCLC (clinical stage IVA or IVB) or recurrent NSCLC (per Version 8 of the International Association for the Study of Lung Cancer [IASLC] Staging Manual in Thoracic Oncology), not amenable to curative surgery or radiotherapy.
6. The tumour harbors at least 1 of the 4 uncommon EGFR mutations (G719X/L861Q/S768I/T790M), either alone or in combination, which not include other EGFR mutations including ex19del /L858R, assessed by one of ARMS, Super-ARMS or NGS analysis on the basis of tumour tissue or plasma testing from accredited laboratories approved by the Chinese regulatory authority.
7. Participants must be considered suitable by investigator and about to receive standard of care which composed of pemetrexed plus carboplatin or cisplatin for 4 to 6 cycles followed by pemetrexed maintenance.
8. Participants must have untreated advanced NSCLC not amenable to curative surgery or radiotherapy. Prior adjuvant and neo-adjuvant therapies (chemotherapy, radiotherapy, immunotherapy, biologic therapy, investigational agents), or definitive radiation/chemoradiation with or without regimens including immunotherapy, biologic therapy, investigational agents, are permitted as long as treatment was completed at least 6 months prior to the development of recurrent disease.
9. Stable CNS metastases participants will be allowed.
10. ECOG/WHO PS of 0 to 1 at screening with no clinically significant deterioration in the previous 2 weeks.
11. Life expectancy >12 weeks at Day 1.
12. At least 1 lesion, not previously irradiated that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have a short axis of ≥15 mm) with CT or MRI, and that is suitable for accurate repeated measurements. If only 1 measurable lesion exists, it is acceptable to be used (as a target lesion) as long as it has not been previously irradiated and as long as it has not been biopsied within 14 days of the baseline tumour assessment scans.
13. Female must be using highly effective contraceptive measures, must not be breast feeding, and must have a negative pregnancy test prior to first dose of study intervention or must have evidence of non-child-bearing potential by fulfilling 1 of the following criteria at screening:

    * Post-menopausal, defined as more than 50 years of age and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
    * Women under 50 years old would be considered as postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution
    * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation. Further information is available in Appendix E (Definition of Women of Childbearing Potential and Acceptable Contraceptive Methods).
14. Male participants must be willing to use barrier contraception.

Exclusion Criteria:

1.Spinal cord compression; symptomatic and unstable brain metastases, except for those participants who have completed definitive therapy, are not on steroids, and have a stable neurological status for at least 2 weeks after completion of the definitive therapy and steroids. Participants with asymptomatic brain metastases can be eligible for inclusion if in the opinion of the Investigator immediate definitive treatment is not indicated.

2 Past medical history of ILD, drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD.

3 Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the participant to participate in the trial or which would jeopardize compliance with the protocol, or active infection including any patients receiving treatment for infection but not limited to hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.

4.Any of the following cardiac criteria:

* Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine-derived QTcF value;
* Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG; eg, complete left bundle branch block, third-degree heart block, second-degree heart block;
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as electrolyte abnormalities including serum/plasma potassium*, magnesium* and calcium* below the lower limit of normal (LLN), heart failure, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes.

  5.Inadequate bone marrow or organ function reserve as demonstrated by any of the following laboratory values:
* Absolute neutrophil count below the LLN *
* Platelet count below the LLN*
* Hemoglobin <90 g/L* *The use of granulocyte colony stimulating factor support, platelet transfusion and blood transfusions to meet these criteria is not permitted.
* ALT >2.5 x the upper limit of normal (ULN) if no demonstrable liver metastases or >5 x ULN in the presence of liver metastases
* AST >2.5 x ULN if no demonstrable liver metastases or >5 x ULN in the presence of liver metastases
* Total bilirubin >1.5 x ULN if no liver metastases or >3 x ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases
* Creatinine clearance <60 mL/min calculated by Cockcroft and Gault equation (refer to Appendix G for appropriate calculation) 6.Any concurrent and/or other active malignancy that has required treatment within 2 years of first dose of study intervention (osimertinib, carboplatin and pemetrexed).

  7 Any unresolved toxicities from prior therapy (eg, adjuvant chemotherapy) greater than CTCAE Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy. 8 Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib.

  9.Prior treatment with any systemic anti-cancer therapy for advanced NSCLC not amenable to curative surgery or radiation including chemotherapy, biologic therapy, immunotherapy, or any investigational drug. Prior adjuvant and neo-adjuvant therapies (chemotherapy, radiotherapy, biologic therapy, investigational agents), or definitive radiation/chemoradiation with or without regimens including biologic therapies, investigational agents are permitted as long as treatment was completed at least 6 months prior to the development of recurrent disease.

  10.Prior treatment with an EGFR-TKI or immune-oncology (IO) therapy. 11.Major surgery within 4 weeks of the first dose of study intervention. Procedures such as placement of vascular access, biopsy via mediastinoscopy or biopsy via video assisted thoracoscopic surgery (VATS) are permitted.

  12.Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study intervention.

  13.Current use of (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of cytochrome P450 (CYP) 3A4 (at least 3 weeks prior) (Appendix F). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.

  14.Participation in another clinical study with an investigational product during the 4 weeks prior to Day 1. Participants in the follow-up period of an interventional study are permitted.

  15.Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and staff at the study site).

  16.Judgment by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.

  17.Previously enrolled in the present study. 18.Currently pregnant (confirmed with positive pregnancy test) or breast-feeding.

  19.History of hypersensitivity to active or inactive excipients of study intervention or drugs with a similar chemical structure or class to study intervention.

  20.In addition, the following conditions are considered criteria for exclusion:
* Prior allogeneic bone marrow transplant
* Non-leukocyte depleted whole blood transfusion within 120 days of genetic sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, Doctor, Principal Investigator — West China Hospital
Locations (6):
- China (6):
  - Research Site, Chengdu
  - Research Site, Harbin
  - Research Site, Mianyang
  - Research Site, Nanchong
  - Research Site, Yibin
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161C00017&attachmentIdentifier=6f77a587-93ed-43f5-ab9e-fa19f3b8c9cc&fileName=5._D5161C00017_Clinical_Study_Protocol_version_v1.0_EN_1_Redacted_pdfa.pdf&versionIdentifier=
- See also: Redacted Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161C00017&attachmentIdentifier=16aba642-fe81-4b02-b42c-4fd9b6dbb301&fileName=D5161C00017-SAP-V1.0_1_Redacted-pdfa.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161C00017&attachmentIdentifier=371d721b-970f-4318-a920-a6f3e6dc91f3&fileName=MINOVA_CSR_(1)_Redacted_pdfa.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 subjects enrolled in the study in total.
Groups:
- Osimertinib Plus Standard Chemotherapy: Dose Formulation: tablet； Dosage Level(s): osimertinib 80 mg QD for oral administration; Dosage formulation, dose reduction:40 mg QD for oral administration
Period: Overall Study
Arm/Group | Osimertinib Plus Standard Chemotherapy
Started (19 January 2022) | 4
Completed (9 March 2023) | 0
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Osimertinib Plus Standard Chemotherapy Single-arm: Dose Formulation: tablet； Dosage Level(s): osimertinib 80 mg QD for oral administration; Dosage formulation, dose reduction:40 mg QD for oral administration
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 4
Age, Customized [Count of Participants; unit: Participants]
  18-130 | 4
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female and male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not collected | 4

OUTCOME MEASURES:

1. Primary Outcome: ORR
Description: ORR (objective response rate) defined as the percentage of participants who achieved a complete response (CR) or partial response (PR) as their best overall response based on Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 as assessed by the investigator
Time Frame: Due to study early terminated, actual time frame is up to 24 weeks.
Population: All enrolled participants who have received at least 1 dose of study intervention (osimertinib).
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 4
Percentage of Patients | 75.0 [19.4 to 99.4]

2. Secondary Outcome: PFS
Description: PFS (Progression-free survival) will be defined as the time from first dose of study intervention until progression per RECIST 1.1 as assessed by the investigator or death due to any cause prior to PD (progressive disease).
Time Frame: Due to study early terminated, actual time frame is up to approximately 12 months.
Population: All enrolled participants who have received at least 1 dose of study intervention (osimertinib).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 4
Months | NA [3.29 to NA] — Median and upper confidence limit were not reached due to an insufficient number of participants with events.

3. Secondary Outcome: OS
Description: OS (Overall survival) is defined as the time from the first dose of treatment to the date of death, regardless of the actual cause of the subject's death. For participants who are still alive at the time of data analysis or who are lost to follow up, OS will be right-censored at the last recorded date that the participant is known to be alive prior to or at the data cut-off date for the analysis.
Time Frame: Due to study early terminated, actual time frame is up to approximately 13 months.
Population: All enrolled participants who have received at least 1 dose of study intervention (osimertinib).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 4
Months | NA [3.94 to NA] — Median and upper confidence limit were not reached due to an insufficient number of participants with events.

4. Secondary Outcome: DoR
Description: DoR (Duration of response) is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression. The end of response should coincide with the date of progression or death from any cause used for the PFS endpoint. The time of the initial response will be defined as the latest of the dates contributing toward the first visit response of PR or CR. If a participant does not progress following a response, then his/her duration of response will use the PFS censoring time as the end point for their DoR calculation.
Time Frame: Due to study early terminated, actual time frame is up to approximately 12 months.
Population: All enrolled participants who have received at least 1 dose of study intervention (osimertinib) with response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 3
Months | NA [NA to NA] — Median, lower and upper confidence limit were not reached due to an insufficient number of participants with events.

5. Secondary Outcome: Depth of Response (Best Absolute Change in Target Lesion Tumour Size From Baseline)
Description: Depth of response (ie, tumour shrinkage / change in tumour size) by Investigator is defined as the relative change in the sum of the longest diameters of RECIST target lesions at the nadir in the absence of NLs (new lesions) or progression of NTLs (non-target lesions) when compared to baseline. The best absolute change in target lesion tumour size from baseline will be summarized using descriptive statistics. The best change in tumour size will include all assessments prior to progression or start of subsequent anti-cancer therapy.
Time Frame: Due to study early terminated, actual time frame is up to approximately 12 months.
Population: All enrolled participants who have received at least 1 dose of study intervention (osimertinib) with response.
Measure: Median (Full Range); unit: mm
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 3
mm | 47.50 [5.16 to 61.60]

6. Secondary Outcome: DCR
Description: DCR (disease control rate) is defined as the percentage of subjects who have a best overall response of CR or PR or SD (stable disease) by RECIST 1.1 as assessed by the Investigator. For participants with a best overall response of SD, a RECIST assessment of SD must have been observed at least 6 weeks following enrolment to be included in the numerator of the calculation for disease control rate. This is to enable sufficient follow-up to establish SD.
Time Frame: Due to study early terminated, actual time frame is up to approximately 12 months.
Population: All enrolled participants who have received at least 1 dose of study intervention (osimertinib).
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 4
Percentage of patients | 100 [39.8 to 100]

7. Secondary Outcome: TTF
Description: Time to treatment failure (TTF) or death is defined as defined as the time from first dose of study intervention (osimertinib) to earlier of the date of last study intervention administration or death due to any cause. Any participant not known to have permanently discontinued study intervention and not known to have died at the time of the analysis will be censored at the last known time on which the participant was known to be alive. Kaplan-Meier method will be used to estimate the median TTF and its 95% confidence interval.
Time Frame: Due to study early terminated, actual time frame is up to approximately 13 months.
Population: All enrolled participants who have received at least 1 dose of study intervention (osimertinib).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 4
Months | NA [3.29 to NA] — Median and upper confidence limit were not reached due to an insufficient number of participants with events.

8. Secondary Outcome: TFST
Description: Time to first subsequent therapy (TFST) or death is defined as the time from first dose of study intervention to the earlier of the date of anti-cancer therapy (except cisplatin or carboplatin or pemetrexed) start date following study intervention discontinuation or death due to any cause. Any participant not known to have had a subsequent therapy or not known to have died at the time of the analysis will be censored at the last known time to have not received subsequent therapy. Kaplan-Meier method will be used to estimate the median TFST and its 95% confidence interval.
Time Frame: Due to study early terminated, actual time frame is up to approximately 13 months.
Population: All enrolled participants who have received at least 1 dose of study intervention (osimertinib).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 4
Months | NA [3.94 to NA] — Median and upper confidence limit were not reached due to an insufficient number of participants with events.

9. Secondary Outcome: Depth of Response (Best Percentage Change in Target Lesion Tumour Size From Baseline)
Description: Depth of response (ie, tumour shrinkage / change in tumour size) by Investigator is defined as the relative change in the sum of the longest diameters of RECIST target lesions at the nadir in the absence of NLs or progression of NTLs when compared to baseline. Best percentage change in target lesion tumour size from baseline will be summarized using descriptive statistics. The best change in tumour size will include all assessments prior to progression or start of subsequent anti-cancer therapy.
Time Frame: Due to study early terminated, actual time frame is up to approximately 12 months.
Population: All enrolled participants who have received at least 1 dose of study intervention (osimertinib) with response.
Measure: Median (Full Range); unit: percentage change in tumour size
Arm/Group | Osimertinib Plus Standard Chemotherapy Single-arm
Number analyzed (Participants) | 3
percentage change in tumour size | 53.61 [40.57 to 78.67]

ADVERSE EVENTS:
Time Frame: From time of signature of informed consent form until 28 days after last dose of study intervention or until the end of study, whichever occurs earlier, up to 13.7 months when study terminated.
Description: The study was terminated, statistical analyses were not performed.
Arm/Group | Osimertinib Plus Standard Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib Plus Standard Chemotherapy (N=4)
Abdominal pain upper (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Hepatobiliary disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 3
Arrhythmia (Cardiac disorders) | 1
Aspartate aminotransferase increased (Hepatobiliary disorders) | 2
Asthenia (General disorders) | 1
Blood lactate dehydrogenase increased (Hepatobiliary disorders) | 1
Constipation (Gastrointestinal disorders) | 1
COVID-19 (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Gamma-glutamyltransferase increased (Hepatobiliary disorders) | 1
Head discomfort (Nervous system disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Malaise (General disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 2
Pain (General disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 2
Pneumonia (Infections and infestations) | 1
Proteinuria (Renal and urinary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell count decreased (Blood and lymphatic system disorders) | 3

LIMITATIONS AND CAVEATS:
Enrollment to study D5161C00017 was terminated prior to completion of the study due to the delay in study enrollment. Due to the early termination of the study, only 4 participants (of the planned 35 participants) received study intervention and data collection for these participants was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT05215951/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT05215951/SAP_001.pdf